CLINICAL TRIAL: NCT01805999
Title: Effect of Ispaghula on Colonic Water Content
Brief Title: Ispaghula and Colonic Water Content
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H13122012SCS
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Healthy
Keywords: Ispaghula; Gastrointestinal physiology; Gastrointestinal response to sugars; MRI; gastrointestinal; stomach; small bowel; colon
MeSH Terms: interventions — Psyllium

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 7 g Ispaghula (Experimental): Volunteer will take 7 g of ispaghula 3 times daily for one week
  Interventions: Dietary Supplement: 7 g Ispaghula
- 7 g placebo (Placebo Comparator): Volunteer will take 7 g of a placebo 3 times a day for one week
  Interventions: Dietary Supplement: 7 g placebo
- 3.5g ispaghula + 3.5 g placebo (Active Comparator): Volunteers will take 3.5 g of ispaghula with 3.5 g placebo 3 times daily for one week
  Interventions: Dietary Supplement: 3.5g Ispaghula + 3.5 g placebo

INTERVENTIONS:
Dietary Supplement: 7 g Ispaghula
  Other Names: Metamucil
  Arms: 7 g Ispaghula
Dietary Supplement: 7 g placebo
  Arms: 7 g placebo
Dietary Supplement: 3.5g Ispaghula + 3.5 g placebo
  Arms: 3.5g ispaghula + 3.5 g placebo

SUMMARY:
Chronic constipation is a phenomenon which affects nearly 20% of the population worldwide. Bulking agents such as ispaghula are used as treatments, but only half of the patients are satisfied with the treatment. This highlights a need for better treatment options, which requires a deeper understanding of the gastrointestinal fate of the products. The GI MRI Research group at the University of Nottingham has been developing new, non-invasive magnetic resonance imaging (MRI) techniques to image the gastrointestinal tract. In collaboration with Ironwood Pharmaceuticals, the investigators now want to understand the gastrointestinal fate of an ispaghula treatment, and also to improve the understanding of MRI parameters when they are applied to the colon.

DETAILED DESCRIPTION:
The Rome III diagnostic criteria for constipation must include two or more of the following symptoms > 25 % of the time: straining, hard or lumpy stools, sense of incomplete evacuation, sensation of anorectal obstruction/blockage, the use of manual manoeuvres to facilitate defecation and fewer than 3 defecations per week. Treatments include osmotic laxatives such as polyethylene glycol and lactulose, stimulant laxatives such as bisacodyl, secretagogues like sodium docusate, and bulking agents such as psyllium.

A better understanding of the modes of action of these drugs is required, in order to provide better treatment for chronic constipation. This is somewhat challenging; partly because techniques available to study intestinal contents are limited, and some are unpleasant for the patients. The GI MRI group at the University of Nottingham has recently developed a non-invasive, patient friendly MRI technique for studying the colon. The technique allows assessment of colonic volumes, the response to meals, motility of the colon and transit time of ingested meals. This technique has been used to demonstrate the laxative effect of mannitol and its subsequent reversal with loperamide.

Using MRI, water provides a bright image on T2-weighted images in the small bowel, but the signal is rapidly lost once it reaches the colon. Pilot studies suggest that ispaghula; which is highly hygroscopic and can form a 1.5% gel with water, is able to maintain water in a form which produces bright images on T2-weighted scanning of the colon. The GI MRI group now want to confirm this pilot data by performing a placebo controlled trial of ispaghula husk in healthy volunteers, with the aim of further understanding the mode of action of bulking agents and further improve understanding of MRI parameters when applied to the colon. The aims will be achieved by performing a dose-finding mechanistic study in healthy volunteers, assessing their response to a test meal while taking either placebo, or 2 different doses of ispaghula. Stools will be collected, assessed for water content and compared to water content assessed from T2 weighted MRI. The studies will validate the current technique, optimise current MRI parameters and provide insights into the modes of action of ispaghula.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy; free from GI disorders, aged 18 and 65 years of age
* Male or female
* Body mass index (BMI) between 18.0 and 30.0 kg m-2
* Suitable for MRI scanning (eg absence of metal implants, infusion pumps and pacemakers as assessed by the MRI safety questionnaire
* No known gastrointestinal disease
* Not currently smoking
* No strenuous exercise greater than 10 hours per week
* No consumption of more than 21 units of alcohol in a typical week
* No reported participation in another nutritional or biomedical trial 3 months before the pre-study examination or during the study.

Exclusion Criteria:

* Inability to discontinue medication likely to alter GI transit
* Antibiotics in the 3 weeks before the pre-study examination
* Pre-existing condition making the need for antibiotics likely during the study
* Previous gastrointestinal surgery (excluding cholecystectomy and appendectomy)
* Known inflammatory bowel disease; coeliac disease
* Subjects considered by the investigator unlikely to comply with study protocol
* Regular (>3 times/week) use of Probiotics in the 3 weeks prior to, or during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
ascending colon free water content (ACWC) | 0 - 360 minutes
  An assessment of the volume of water in the ascending colon, as obtained from MR images

SECONDARY OUTCOMES:
Ascending, transverse and descending colon volumes | 0 - 360 minutes
  The volumes of each region of the colon will be determined by segmenting MR images
Geometric centres (GC) 24 and 48 hours | t = 24 hours and t = 48 hours
  The geometric centres of 5 transit marker pills will be determined at 24 and 48 hours after ingestion
Small bowel water content | 0 - 360 minutes
  The volume of water in the small bowel will be evaluated from the MR images over the study day
Gastric emptying | 0 - 360 minutes
  The rate of gastric emptying throughout the study day will be determined from MR images

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, MD, FRCP, Study Chair — University of Nottingham; Jeffrey Johnston, MD, FACP, Study Director — Ironwood Pharmaceuticals, Inc.; Luca Marciani, Laurea, PhD, Principal Investigator — University of Nottingham; Kathryn Murray, PhD, Principal Investigator — University of Nottingham; Giles Major, MB BChir, Principal Investigator — University of Nottiingham; Ching Lam, MB BCh, Principal Investigator — University of Nottingham; Caroline Hoad, PhD, Principal Investigator — University of Nottingham; Penny Gowland, PhD, Principal Investigator — University of Nottingham
Locations (1):
- NDD BRU and Sir Peter Mansfield Magnetic Resonance Centre, Nottingham, Nottinghamshire, United Kingdom